CLINICAL TRIAL: NCT03471689
Title: Multisensory Integration and Pain Perception
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00046662
Record Dates: First submitted 2018-03-12; First posted 2018-03-20 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Pain; Regulation, Self
Keywords: Multimodal; Pain perception; Regulation; Mindfulness
MeSH Terms: conditions — Pain; Self-Control | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental)
  Interventions: Behavioral: Mindfulness meditation
- Positive reappraisal (Active Comparator)
  Interventions: Behavioral: Positive reappraisal

INTERVENTIONS:
Behavioral: Mindfulness meditation — Participants will be trained to use mindfulness meditation to reduce pain perception.
  Arms: Mindfulness
Behavioral: Positive reappraisal — Participants will be trained to use positive reappraisal to reduce pain perception.
  Arms: Positive reappraisal

SUMMARY:
Pain is a predominant disruption of well-being among humans. Feeling pain is a multimodal sensory experience where information is collected and processed from various senses such as sight and touch. Because pain is complex, variable, and experienced differently by each individual, finding more accessible and practical treatments for pain are necessary. Mindfulness meditation (MM) aims to reduce pain by directing focus to perceive thoughts through non-judgmental awareness. Positive reappraisal (PR) is a possible cognitive pain treatment that focuses on changing the meaning of stressful or negative events into positive, benign, valuable, or beneficial. When a stressful event, such as experiencing pain, is positively reappraised, the individual recognizes and engages with the feeling of stress produced by the event and intentionally looks for benefits that change the feeling from negative to positive. The focus of this study is to examine the effect of different cognitive techniques on multimodal innocuous and noxious stimuli. Visual and tactile noxious stimuli will be administered to determine how visual cue integrate to form and modulate the subjective experience of pain. The study team postulates that mindfulness meditation and positive reappraisal will significantly reduce pain in response to multimodal stimulus (visual cue + noxious heat) when compared to a non-manipulation control condition. These findings will be utilized to better understand the multidimensional mechanisms supporting nociception and the cognitive modulation of pain.

ELIGIBILITY:
Inclusion Criteria:

* Native/fluent English speaker
* Ability to understand/willingness to sign consent form

Exclusion Criteria:

* Chronic pain
* Cardiac medications
* Diagnosis of mental illness or personality disorder
* Diagnosis of heart or lung conditions/hyper tension
* Taking psychiatric medications

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Psychophysical Assessment of Pain | throughout study completion, up to 2 hours
  Pain intensity and unpleasantness ratings will be assessed with the Visual Analogue Scale (VAS). If the participant states that he or she "is in no pain" or the pain "is not at all unpleasant," a rating of 0 will be recorded for pain intensity and unpleasantness, respectively. The maximum rating of "10" will designate the "most intense pain imaginable/the most unpleasant pain imaginable".
Assessment of Physiologic Measurements | throughout study completion, up to 2 hours
  Participants may be fitted with electrocardiography (ECG) sensors and a respiratory belt that is placed around the participant's chest. Subjects may also be fitted with sensors that measure electrodermal activity. All physiological activity will be recorded at a rate of 1 kHz and will be processed with an integrated software system. Respiratory rate will be calculated in breaths per minute. ECG sensors will be placed on the lower right and left ribs of the participant. Respiration belt will be attached to the upper chest, and two 6 mm Ag/AgCl skin conductance electrodes will be placed on the distal phalanges of the first and second fingers of the non-dominant hand. Higher scores reflect more physiological arousal to pain stimuli.
Freiburg Mindfulness Inventory (FMI) (Short Form) | throughout study completion, up to 2 hours
  This 14-item form assesses self- attributed mindfulness. The inventory is composed of 14 items that use a 1 to 4 Likert scale. Obtaining a higher score represents higher mindfulness.
Ways of Coping Scale (WOCS-PR; Positive Reappraisal Subscale) | throughout study completion, up to 2 hours
  The 7-item form assesses levels of positive reappraisal. The WOCS- Positive Reappraisal Subscale has a total of seven questions. It uses a Likert scale ranging from 0 to 3 and asks the participant to think of a specific stressful situation. High scores on the PR subscale represent frequent use by the individual of positive reappraisal for stressful events.
State Anxiety Inventory (SAI) | throughout study completion, up to 2 hours
  This 20-item scale is commonly used to measure state anxiety and has internal consistency, construct validity, and test-retest reliability. A score between 20 and 80 is given, with higher scores representing higher levels of anxiety.
Pain Catastrophizing Scale (PCS) | throughout study completion, up to 2 hours
  This 13-item form assesses rumination, magnification, and helplessness, attributes used in the literature to define pain catastrophizing. Each item is given a score from 0 to 4. The total scores range from 0 to 52, with higher ratings representing higher levels of catastrophic thinking.
Positive and Negative Affective Scale (PANAS) | throughout study completion, up to 2 hours
  This scale measures general affective states by assessing a subject's experience of 20 different emotions. This scale is scored on a 5-point scale, with higher scores for the positive questions representing higher levels of positive affect, and higher scores for the negative questions representing higher levels of negative affect.
Beck Depression Inventory (BDI) | throughout study completion, up to 2 hours
  This scale is a 21-question multiple-choice self-report inventory for measuring the severity of depression, and it has internal consistency, construct validity, and test-retest reliability. There is a total of 21 questions with a Likert scale ranging from 0 to 3. Higher scores represent higher levels of depression.
Perceived Stress Scale (PSS) | throughout study completion, up to 2 hours
  This is a psychological instrument for measuring participant's perception of stress. It has internal consistency, construct validity, and test-retest reliability. There is a total of 10 questions with higher scores denoting higher levels of perceived stress.
VAS of Analgesia | throughout study completion, up to 2 hours
  Participants will be asked to indicate, by using the visual analog scale, how much pain they will expect to experience. If the participant states that he or she "will experience no pain" or the pain "will not be unpleasant," a rating of 0 will be recorded for pain intensity and unpleasantness, respectively. The maximum rating of "10" will designate the "most intense pain imaginable/the most unpleasant pain imaginable".
VAS of Political Affiliation | throughout study completion, up to 2 hours
  Using the VAS, participants will indicate where in the political spectrum they identify. Participants will be instructed that the right side of the VAS corresponds to conservatism while the left corresponds to liberalism. Participants will move the sliding scale on the VAS to the location corresponding to their political affiliation.
VAS of Stress | throughout study completion, up to 2 hours
  Participants will indicate with the VAS how stressed, from a scale of 0-10, they are at the present moment. A rating of 0 will be recorded for "no stress" while a rating of 10 will be recorded for "highest" stress possible.
Valence Ratings for Images | throughout study completion, up to 2 hours
  : Participants for phase one will rate the images based on the International Affective Picture System (IAPS) valence ratings. The ratings will use a Likert scale ranging from 1 (low pleasantness) to 9 (high pleasantness). After the participants look at the image for 2 seconds, they will be asked to rate level of pleasantness in less than 5 seconds based on the immediate feeling experienced while viewing the image.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Waugh, PhD, Principal Investigator — Wake Forest University; Fadel Zeidan, PhD, Principal Investigator — Wake Forest University Health Science
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No